CLINICAL TRIAL: NCT06016790
Title: Scientific Research on Exploring a Breast Cancer Early Screening Model Using cfDNA Multi-omics Liquid Biopsy Technology Based on Deep Learning
Brief Title: Exploring a Breast Cancer Early Screening Model Based on cfDNA
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: OmixScience Institute (Unknown)
Responsible Party: Principal Investigator, Ni Chao, Associate Chief Physician of Breast Surgery, Second Affiliated Hospital, School of Medicine, Zhejiang University
Other Study IDs: ZE-OMIX-001
Record Dates: First submitted 2023-08-22; First posted 2023-08-30 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Breast Fibroadenoma; Breast Hypoplasia
Keywords: cfDNA; Deep learning
MeSH Terms: conditions — Breast Neoplasms; Fibroadenoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Biospecimen Retention: Samples With DNA — peripheral venous blood with cfDNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- the cancer group: 503 cases of early breast cancer
  Interventions: Genetic: cfDNA sequencing
- the benign control group: 289 cases of control group
  Interventions: Genetic: cfDNA sequencing

INTERVENTIONS:
Genetic: cfDNA sequencing — Multi-omics sequencing of cfDNA in peripheral venous blood.

SUMMARY:
The goal of this observational study is to use cfDNA multi-omics technology to explore a new breast cancer early detection model to improve the accuracy of early diagnosis in breast cancer patients. The main questions it aims to answer are:

* Evaluate the sensitivity and specificity of the early detection model for breast cancer screening
* Evaluate participants' TeFei™ score Participants will be collected peripheral venous blood before surgery or systemic treatment. The blood will then be sent to the collaboration company for sequencing. The collaboration company will analyze the sequencing results and build a cfDNA multi-omics signature library. Finally, the collaboration company will use deep learning algorithms to train and optimize the feature library.

Researchers will compare the cancer group with a benign control group to determine the model's effectiveness in differentiating between them.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years old and ≤70 years old;
2. Plasma of the participant can be obtained;
3. Willing to sign the informed consent;
4. Meet one of the following criteria:

4.1)Patients diagnosed with invasive breast cancer or carcinoma in situ of the breast for the first time; 4.2)Patients with breast fibroma or breast adenosis and breast fibrocystic hyperplasia;

Exclusion Criteria:

In any of the following situations, subjects should not participate in the trial:

1. Pregnant or lactating;
2. Unable to obtain the participant's plasma;
3. Patients with other types of malignant tumors diagnosed by pathology within 5 years before enrollment;
4. The patients had suspected imaging (B-ultrasound, CT, etc.) of other malignant tumors within the past 1 year after enrollment, but no pathological confirmation;
5. Received any blood product transfusion in the past 30 days;
6. Participants considered by the investigator to be inappropriate to participate in this research-type clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients and patients with benign breast diseases.
Sampling Method: Non-Probability Sample
Enrollment: 839 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Evaluate the sensitivity and specificity of the early detection model for breast cancer screening | 1 year from enrollment
  Peripheral blood samples were collected during routine physical examinations for healthy volunteers and prior to surgery for cancer patients. The blood samples were drawn and placed into cfDNA preservation tubes (Ardent BioMed, Guangdong, China, Cat. # BY10240301). After collection, the fresh blood was subjected to an initial centrifugation at 1,600 × g for 10 minutes at 4°C, allowing the plasma supernatant to be carefully separated via pipetting. This plasma was then centrifuged again at 16,000 × g for 10 minutes at 4°C to remove any residual debris. The resulting plasma supernatant was then carefully collected and stored at -80°C. The preserved plasma samples were subsequently transported on dry ice to the central laboratory at OmixScience Research Institute (Hangzhou, China).

SECONDARY OUTCOMES:
Evaluate participants' TeFei™ score | 60 days
  This test is based on the expression level of key genes in the cfDNA tumor of the participant's blood sample, and the relative expression level of these genes is calculated to obtain a score. This score is called the TeFei™ Score and usually ranges from 0 to 100, with a higher score indicating a higher tumor burden in the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Chao Ni, Principal Investigator — Second Affiliated Hospital of Zhejiang University School of Medicine
Locations (8):
- China (8):
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu, Anhui
  - Affiliated Hangzhou First People's Hospital ,Westlake University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital Affiliated With Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Wenhui Community Health Service center, Gongshu district, Hangzhou city, Hangzhou, Zhejiang
  - Women's Hospital School Of Medicine Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Provincial Hospital Of Traditional Chinese Medicine, Hangzhou, Zhejiang
  - Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No
Because the database is related to the products of the cooperative company, in order to protect the intellectual property rights of the cooperative company, IPD will not be shared.

REFERENCES:
- [Background] Mathios D, Johansen JS, Cristiano S, Medina JE, Phallen J, Larsen KR, Bruhm DC, Niknafs N, Ferreira L, Adleff V, Chiao JY, Leal A, Noe M, White JR, Arun AS, Hruban C, Annapragada AV, Jensen SO, Orntoft MW, Madsen AH, Carvalho B, de Wit M, Carey J, Dracopoli NC, Maddala T, Fang KC, Hartman AR, Forde PM, Anagnostou V, Brahmer JR, Fijneman RJA, Nielsen HJ, Meijer GA, Andersen CL, Mellemgaard A, Bojesen SE, Scharpf RB, Velculescu VE. Detection and characterization of lung cancer using cell-free DNA fragmentomes. Nat Commun. 2021 Aug 20;12(1):5060. doi: 10.1038/s41467-021-24994-w. PMID 34417454
- See also: Freenome, a privately held biotech company, announced the completion of enrollment for PREEMPT CRC, the company's large, prospective study to validate its blood test for colorectal cancer (CRC) screening among average-risk adults. — http://www.freenome.com/largest-clinical-study-validating-a-blood-based-colorectal-screening-test-completes-enrollment